CLINICAL TRIAL: NCT01462604
Title: PROACTYVE Pilot:Pilot Study of Patient's Adherence to TYKERB™/TYVERB™+Capecitabine in Metastatic Breast Cancer-Observation of Patient Adherence and Evaluation of Predictive Factors for Patient Adherence After Providing Educational Programme
Brief Title: Pilot Study of Patient's Adherence to TYKERB™/TYVERB™ + Capecitabine in Metastatic Breast Cancer
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 115553
Record Dates: First submitted 2011-09-21; First posted 2011-10-31 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HER2 overexpressing metastatic or advanced breast cancer pts
  Interventions: Other: non-drug intervention educational programme

INTERVENTIONS:
Other: non-drug intervention educational programme — educational programme

SUMMARY:
This is a 6-week, single arm, pilot study to test the study procedure, educational materials, and measurement instruments for the educational intervention in HER2 overexpressing metastatic or advanced breast cancer patients

DETAILED DESCRIPTION:
Approximately 60 subjects with HER2+ metastatic or advanced breast cancer who meet the inclusion/exclusion criteria will be enrolled into the study. All subjects will receive education intervention for 6 weeks including education on Day 0, follow-up phone calls on Day 1 and Day 7, reminder phone calls before Week 3 and 6 visit and telephone hot line number.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent;
2. Female outpatient aged 18 years or older;
3. Subjects must be about to begin their initial treatment with lapatinib + capecitabine for HER2+ metastatic or advanced breast cancer according to physician's clinical judgement as per local prescribing information
4. Subjects must be literate, be able to read, understand and write local language.

Exclusion Criteria:

1. Women who is participating in any other interventional clinical trials concurrently;
2. Women who is already taking or had taken lapatinib + capecitabine regimen prior to the enrollment;
3. Primary lesions that are not of breast origin.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women older than 18 years old with metastatic or advanced breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2011-11-23; Primary Completion 2013-01-01 (Actual); Study Completion 2013-01-24 (Actual)

PRIMARY OUTCOMES:
Subject recruitment and retention in the study | upto week 6
  Assess the feasibility of recruitment and retention of subjects into the education program
Adherence at Week 3 and Week 6 (MARS-6) and persistence at Week 6 | week 3 & 6
  Pilot test tools to measure subject adherence to the lapatinib + capecitabine regimen, assess persistence and describe these outcomes
Patient knowledge, attitude and beliefs about the regimen | Day 0, Week 3 and Week 6
  Pilot test tools to measure subject knowledge, attitudes, and beliefs about the lapatinib + capecitabine regimen and describe these outcomes
Acceptability of study procedures and educational materials at Week 6 | week 6
  Evaluate the implementation and acceptability of the education materials and study procedures

SECONDARY OUTCOMES:
Serious adverse events and adverse events up to 6 weeks | upto week 6
  Safety during education intervention

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- Hong Kong (2):
  - GSK Investigational Site, Pokfulam
  - GSK Investigational Site, Shatin
- Pakistan (2):
  - GSK Investigational Site, Karachi
  - GSK Investigational Site, Lahore
- GSK Investigational Site, Singapore, Singapore
- GSK Investigational Site, Seoul, South Korea